CLINICAL TRIAL: NCT02720744
Title: A Double-blind, Randomized, Placebo Controlled, Two Arm Multi-center Study to Assess the Efficacy and Safety of a Once Nightly Formulation of Sodium Oxybate for Extended-Release Oral Suspension (FT218) for the Treatment of Excessive Daytime Sleepiness and Cataplexy in Subjects With Narcolepsy
Brief Title: Once-Nightly Sodium Oxybate for Treatment of Excessive Daytime Sleepiness and Cataplexy in Narcolepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avadel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLFT218-1501
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Excessive Daytime Sleepiness; Cataplexy; Narcolepsy
MeSH Terms: conditions — Disorders of Excessive Somnolence; Cataplexy; Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Oxybate (Experimental): Patients will undergo a screening period and will then be titrated to the following once-nightly doses: 4.5 g sodium oxybate, 6.0 g sodium oxybate, 7.5 g sodium oxybate, and 9.0 g sodium oxybate.
  Interventions: Drug: FT218
- Placebo (Placebo Comparator): Patients will undergo a screening period and will then be titrated to the following once-nightly doses: 4.5 g placebo, 6.0 g placebo, 7.5 g placebo, and 9.0 g placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FT218
  Arms: Sodium Oxybate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether once-nightly FT218 is safe and effective for the treatment of excessive daytime sleepiness and cataplexy in subjects with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 16 years of age or older
2. Willing and able to give written informed consent for study participation. For young adults (16 and 17 years old) who have not reached the age of majority they must be capable of giving assent and consent from a legally authorized guardian must be obtained, as required by local laws and regulations
3. Documented evidence of a diagnosis of NT1 (type 1 narcolepsy) or NT2 (type 2 narcolepsy) as, in part, determined by an overnight PSG (polysomnography) and next-day MSLT (maintenance of sleep latency test) with 2 or more SOREMPs (sleep onset REM) with mean sleep latency in the pathological range i.e. < 8 minutes and meeting the NT1 and NT2 as defined by the International Classification of Sleep Disorders -3 criteria.
4. Current continuing presence of EDS (excessive daytime sleepiness) as defined by subject report for the last 3 months and an ESS (Epworth sleepiness scale) > 10
5. For NT1 only, current continuing presence of cataplexy as defined by subject report for the last 3 months
6. Subjects may use concomitant stimulants, but must comply with the following:

   1. They must be on a stable dose of stimulants for at least 3 weeks prior to starting the screening process for this study; AND
   2. They must use the same stimulant regimen throughout the entire study period, including during screening and posttreatment periods
   3. They must discontinue all anti cataplexy drugs
7. Addition inclusion criteria per protocol

Exclusion criteria

1. Any prior use of sodium oxybate is allowed in the study but within the following exclusions:

   1. Previous dosing must have been limited to no more than 4.5g per night
   2. Patient should not have taken sodium oxybate for more than 2 weeks.
   3. All previous dosing must not have occurred within the last year prior to entry to the study.
2. Current use of sodium valproate
3. Any use of the following prohibited medications for the duration of the clinical study:

   1. Anticonvulsants
   2. Clonidine
   3. SSRIs (selective serotonin re-uptake inhibitors) and serotonin and norepinephrine re-uptake inhibitors (SNRIs)
   4. MAOIs (monoamine oxidase inhibitors)
   5. TCAs (tricyclic antidepressants)
   6. Hypnotics
   7. Anxiolytics
   8. Sedating antihistamines
   9. Antipsychotics
   10. Other experimental medications designed to treat narcolepsy, cataplexy or any other condition
4. Treatment with any investigational products within 3 months before study enrollment
5. Any drug known to affect sleep-wake function. Concomitant stimulant use is permitted
6. Additional exclusion criteria per protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (38):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - University Sleep Disorder Center, Auburn, Alabama
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - California Center for Sleep Disorders, Alameda, California
  - Stanford Sleep Medicine, Redwood City, California
  - SDS Clinical Trials Inc, Santa Ana, California
  - Alpine Research Center, Boulder, Colorado
  - Yale-New Haven Hospital's Sleep Medicine Center, North Haven, Connecticut
  - Pulmonary Disease Specialist, PA, Kissimmee, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Sleep Medicine Specialist of South Florida, Miami, Florida
  - NeuroMedical Research Institute/Global Research Holdings, LLC, Panama City, Florida
  - FL Pediatric REsearch Institute, Winter Park, Florida
  - Florida Pulmonary Research Institute LLC, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - OSF Healthcare Saint Francis Medical Center, Peoria, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Norton Clinical Research Group, Louisville, Kentucky
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Northwell Health, New Hyde Park, New York
  - Clinilabs Drug Development Corporation, New York, New York
  - Montefiore Sleep-Wake Disorders Center, The Bronx, New York
  - Research Carolina of Huntersville, Huntersville, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Sleep Management Institute Intrepid Research, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Medical University of South Carolina - Institute of Psychiatry, Charleston, South Carolina
  - SleepMed Of South Carolina, Columbia, South Carolina
  - Sleep and Neurology Consultants, Houston, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
- Australia (6):
  - NHMRC CEntre for Translational Sleep and Circadian Neurobiology, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Melbourne Sleep Disorders Centre, Melbourne, Victoria
- Canada (6):
  - Somni Research Inc. Calgary, Calgary, Alberta
  - Okanagan Clinical Trials Ltd, Kelowna, British Columbia
  - West Parry Sound Health Center, Parry Sound, Ontario
  - Somni Research Inc, Toronto, Ontario
  - Paediatric Sleep Research Inc, Toronto, Ontario
  - CIUSS de Nord-de-I'ile-de- Montreal- Hopital de Sacre-Coeur de Montreal, Montreal, Quebec
- Vseobecna Facultni Nemocnice, Prague, Czechia
- France (3):
  - CHU Michallon, Grenoble
  - Hospital Gui-de-de-Chauliac, Montpellier
  - INSERM - Centre d'Investigation Clinque Hopital Robert Debre, Paris
- Germany (3):
  - Charit Universittsmedizin Berlin, Berlin
  - Hephata Klinik, Schwalmstadt
  - Somni bene GmbH, Schwerin

REFERENCES:
- [Derived] Ortiz LE, Morse AM, Thorpy MJ, Kushida CA, Harsh J, Roth T, Gudeman J, Dauvilliers Y. Once-Nightly Sodium Oxybate Meets American Academy of Sleep Medicine Criteria for Treatment of Narcolepsy. J Sleep Res. 2025 Aug 25:e70189. doi: 10.1111/jsr.70189. Online ahead of print. PMID 40851446
- [Derived] Roth T, Thorpy MJ, Kushida CA, Gudeman J. Efficacy of Once-Nightly Sodium Oxybate in Patients with Narcolepsy: Post Hoc Analyses of Sensitivity, Effect Size, and Numbers Needed to Treat from the Phase 3 REST-ON Trial. CNS Drugs. 2025 Mar;39(Suppl 1):61-70. doi: 10.1007/s40263-025-01160-0. Epub 2025 Mar 20. PMID 40111739
- [Derived] Krahn L, Roy A, Winkelman JW, Morse AM, Gudeman J. Assessing Early Efficacy After Initiation of Once-Nightly Sodium Oxybate (ON-SXB; FT218) in Participants with Narcolepsy Type 1 or 2: A Post Hoc Analysis from the Phase 3 REST-ON Trial. CNS Drugs. 2025 Mar;39(Suppl 1):53-59. doi: 10.1007/s40263-024-01143-7. Epub 2025 Mar 20. PMID 40111738
- [Derived] Dauvilliers Y, Roth T, Bogan R, Thorpy MJ, Morse AM, Roy A, Gudeman J. Efficacy of once-nightly sodium oxybate (FT218) on daytime symptoms in individuals with narcolepsy with or without concomitant alerting agent use: A post hoc analysis from the phase 3 REST-ON trial. Sleep Med. 2024 Dec;124:209-216. doi: 10.1016/j.sleep.2024.09.024. Epub 2024 Sep 17. PMID 39321628
- [Derived] Roth T, Morse AM, Bogan R, Roy A, Gudeman J, Dauvilliers Y. Weight Loss With Once-nightly Sodium Oxybate for the Treatment of Narcolepsy: Analysis From the Phase III Randomized study Evaluating the efficacy and SafeTy of a ONce nightly formulation of sodium oxybate (REST-ON) Trial. Clin Ther. 2024 Oct;46(10):791-798. doi: 10.1016/j.clinthera.2024.07.010. Epub 2024 Aug 16. PMID 39153911
- [Derived] Roth T, Dauvilliers Y, Thorpy MJ, Kushida C, Corser BC, Bogan R, Rosenberg R, Dubow J, Seiden D. Effect of FT218, a Once-Nightly Sodium Oxybate Formulation, on Disrupted Nighttime Sleep in Patients with Narcolepsy: Results from the Randomized Phase III REST-ON Trial. CNS Drugs. 2022 Apr;36(4):377-387. doi: 10.1007/s40263-022-00904-6. Epub 2022 Apr 5. PMID 35380374
- [Derived] Kushida CA, Shapiro CM, Roth T, Thorpy MJ, Corser BC, Ajayi AO, Rosenberg R, Roy A, Seiden D, Dubow J, Dauvilliers Y. Once-nightly sodium oxybate (FT218) demonstrated improvement of symptoms in a phase 3 randomized clinical trial in patients with narcolepsy. Sleep. 2022 Jun 13;45(6):zsab200. doi: 10.1093/sleep/zsab200. PMID 34358324

RESULTS

PARTICIPANT FLOW:
Groups:
- FT218: Patients treated with FT218, once nightly sodium oxybate granules for oral suspension
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | FT218 | Placebo
Started | 107 | 105
Completed | 69 | 79
Not Completed | 38 | 26
Not completed — Protocol Violation | 0 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 2 | 8
Not completed — Adverse Event | 21 | 3
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to follow up | 2 | 0
Not completed — Non Compliance with Investigational Product | 0 | 1
Not completed — Excluded Concomitant Medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FT218 | Placebo | Total
Number analyzed (Participants) | 107 | 105 | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 12 | 21
  Between 18 and 65 years | 97 | 91 | 188
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (10.70) | 31.6 (11.24) | 31.2 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 38 | 30 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 8 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 15 | 36
  White | 80 | 80 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 53 | 116
  Australia | 4 | 7 | 11
  Canada | 28 | 31 | 59
  Czechia | 1 | 1 | 2
  Denmark | 6 | 7 | 13
  France | 3 | 5 | 8
  Netherlands | 1 | 0 | 1
  United Kingdom | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Wakefulness Test (MWT)
Description: Change from Baseline for MWT, which is the mean latency across 5 naps, averaged over the test day
Time Frame: Study Visit 8 at 14 weeks
Population: Maintenance of Wakefulness Test (MWT) Mean Sleep Latency (Minutes) Change from Baseline to the End of the 9.0g Treatment Period - MMRM (mixed model repeat measure) Analysis (mITT Population)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FT218 | Placebo
Number analyzed (Participants) | 68 | 78
minutes | 10.8 (0.96) | 4.7 (0.92)
Statistical Analysis 1: Comparison: FT218 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Each outcome measure for the 9.0 g, 7.5 g, and 6.0 g doses were tested at the 2-sided α level of 0.05; P-values were estimated using an MMRM with change from baseline (or its log transformation); Mean Difference (Net) = 6.13, 95% CI 2-sided [3.52 to 8.75] — Difference from placebo was defined by the FT218 mean value minus placebo value

2. Primary Outcome: Proportion of Patients That Were Very Much Improved or Much Improved on Clinical Global Impression of Improvement as Compared to Screening
Description: The CGI is the clinician's global impression of improvement in daytime sleepiness. For the CGI, a GLIMMIX (generalized linear mixed models) model for binomial data with logit link was used to analyze the categorized CGI response, i.e., the proportions of subjects who were Very Much Improved or Much Improved as compared to Screening
Time Frame: Study Visit 8 at 14 weeks
Population: Clinical Global Impression - Improvement (CGI-I) by the End of 9.0g Treatment Period
Measure: Number; unit: percentage of subjects
Arm/Group | FT218 | Placebo
Number analyzed (Participants) | 69 | 79
percentage of subjects | 72.0 | 31.6
Statistical Analysis 1: Comparison: FT218 vs Placebo; Test type: Superiority; p < 0.001, GLIMMIX model — Each outcome measure for the 9.0 g, 7.5 g, and 6.0 g doses were tested at the 2-sided α level of 0.05; P-values estimated with categorized CGI-Improvement response (very much or much improved versus other category) at the specific visit; Odds Ratio (OR) = 5.56, 95% CI 2-sided [2.76 to 11.23]

3. Primary Outcome: Number of Cataplexy Attacks at Visit 8 (Week 14) as Compared to Baseline
Description: Mean number of cataplexy events recorded on the Sleep and Symptom Daily Diary during the period
Time Frame: Visit 8 - Change from Baseline at 14 Weeks
Population: Mean Weekly Number of Cataplexy Attacks (NCA) of Each Dosing Period, Change from Baseline to the End of 9.0g Treatment Period - MMRM Analysis (NT1 Subjects in mITT Population)
Measure: Mean (Standard Deviation); unit: Cataplexy Attacks
Arm/Group | FT218 | Placebo
Number analyzed (Participants) | 54 | 62
Cataplexy Attacks | -11.5 (0.96) | -4.9 (0.95)
Statistical Analysis 1: Comparison: FT218 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Each outcome measure for the 9.0 g, 7.5 g, and 6.0 g doses were tested at the 2-sided α level of 0.05; P-values were estimated using an MMRM with change from baseline to the end of the respective treatment period; Mean Difference (Net) = -6.65, 95% CI 2-sided [-9.32 to -3.98]

ADVERSE EVENTS:
Time Frame: AE (adverse event) data were obtained at all study visits (scheduled or unscheduled) from the time of the signing of informed consent until seven days after the last dose of study drug, at 14 weeks.
Groups:
- FT218 9g Group; Placebo 9g Group: Patients treated with FT218 who completed the 9g dosing period
Arm/Group | FT218 9g Group | Placebo 9g Group
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/80
Other Adverse Events (participants affected / at risk) | 23/77 | 6/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FT218 9g Group (N=77) | Placebo 9g Group (N=80)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FT218 9g Group (N=77) | Placebo 9g Group (N=80)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0)
Enuresis (Psychiatric disorders) | 7 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Weight Decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02720744/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02720744/SAP_001.pdf